CLINICAL TRIAL: NCT05828095
Title: A Phase 1 Open-label Clinical Trial to Evaluate the Safety and Immunogenicity of Synthetic DNAs Encoding a Native-like HIV Env Trimer and Interleukin-12 (INO-6160), Alone or in a Prime-boost Regimen With 3M-052-AF + Alum Adjuvanted VRC HIV Env Trimer 4571 in Adult Participants Without HIV
Brief Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of Synthetic DNAs Encoding a Native-like HIV Env Trimer and Interleukin-12 (INO-6160), Alone or in a Prime-boost Regimen With 3M-052-AF + Alum Adjuvanted VRC HIV Env Trimer 4571 in Adult Participants Without HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 304
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-07

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — aluminum sulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group #1: INO-6160/ 2.0 mg (Experimental): The dose of INO-6160, 2 mg, will be administered as 2 separate intradermal (ID) injections, one in each arm
  Interventions: Biological: INO-6160, 2 mg
- Group #2: INO-6160/ 2.0 mg with Trimer-4571 / 100 mcg 3M-052-AF (5 mcg) + Alum (500 mcg) (Experimental): The dose of INO-6160, 2 mg, will be administered as 2 separate intradermal (ID) injections, one in each arm.
  The dose of Trimer 4571, 100 mcg, will be administered as 2 injections delivered intramuscularly (IM), one in each arm.
  Interventions: Biological: INO-6160, 2 mg; Biological: Trimer-4571 / 100 mcg 3M-052-AF (5 mcg) + Alum (500 mcg)

INTERVENTIONS:
Biological: INO-6160, 2 mg — ID EP at month 0,1,3 and 6
Biological: Trimer-4571 / 100 mcg 3M-052-AF (5 mcg) + Alum (500 mcg) — IM at month 3 and 6
  Arms: Group #2: INO-6160/ 2.0 mg with Trimer-4571 / 100 mcg 3M-052-AF (5 mcg) + Alum (500 mcg)

SUMMARY:
This is a randomized open-label trial to examine the safety and immunogenicity of INO-6160 (synthetic DNAs encoding a native-like HIV Env Trimer and Interleukin-12), alone or in a prime-boost regimen with VRC HIV Env Trimer 4571 adjuvanted with 3M-052-AF + Alum. The primary hypothesis is that the vaccine regimen will elicit HIV-1 envelope protein-specific binding antibody (Ab) and T-cell responses

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to complete the informed consent process, including an Assessment of Understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of questionnaire items that were answered incorrectly
* 18-55 years old, inclusive, on day of enrollment
* Available for clinic follow-up through the last clinic visit and willing to be contacted 12 months after the last vaccine administration
* Agrees not to enroll in another study of an investigational agent during participation in the trial
* In good general health according to the clinical judgment of the site investigator
* Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator
* Assessed as low risk for HIV acquisition per low risk guidelines, agrees to discuss HIV infection risks, agrees to risk reduction counseling, and agrees to avoid behavior associated with high risk of HIV exposure through the final study visit. Low risk may include persons stably taking PrEP as prescribed for 6 months or longer
* Hemoglobin:

  * ≥ 11.0 g/dL for volunteers who were assigned female sex at birth
  * ≥ 13.0 g/dL for volunteers who were assigned male sex at birth and transgender men who have been on hormone therapy for more than 6 consecutive months
  * ≥ 12.0 g/dL for transgender women who have been on hormone therapy for more than 6 consecutive months
  * For transgender participants who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on their sex assigned at birth
* White blood cell (WBC) count = 2,500-12,000/mm3 (not exclusionary: if count greater than 12,000 with investigation showing general good health and PSRT approval)
* Platelets = 125,000-550,000/mm3
* Alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) based on the institutional normal range
* Serum creatinine ≤ 1.1 x ULN based on the institutional normal range
* Blood pressure in the range of 90 to < 140 mmHg systolic and 50 to < 90 mmHg diastolic
* Negative results for HIV infection by a Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA)
* Negative for anti-Hepatitis C antibodies (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV antibodies are detected
* Negative for Hepatitis B surface antigen
* For a volunteer capable of becoming pregnant:

  * Volunteers who were assigned female sex at birth and are of reproductive potential must agree to use effective means of birth control from at least 21 days prior to enrollment through 8 weeks after their last scheduled fifth vaccination timepoint
  * Has negative β-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment.
  * Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination or in vitro fertilization through 8 weeks after their last scheduled vaccination timepoint

Exclusion Criteria:

* Volunteer who is breast-feeding or pregnant
* Body mass index (BMI). Enrollment of individuals with BMI ≥ 40, whom the site investigator assesses are in good health, may be considered by PSRT on a case-by-case basis
* Diabetes mellitus (DM). Type 2 DM controlled with diet alone, or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well-controlled on diet alone or on hypoglycemic agent(s) may be considered, provided the HgbA1c is ≤8% within the last 6 months (sites may draw these at screening)
* Previous or current recipient of an investigational HIV vaccine (previous placebo recipients are not excluded)
* Congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator such as glucocorticoid use equal to or greater than prednisone 10 mg/day within 3 months prior to enrollment
* Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval
* Receipt of any live attenuated vaccine within 4 weeks prior to enrollment
* ACAM2000 vaccine for Monkeypox received within 30 days prior to enrollment or receipt of study product, or if ACAM2000 received greater than 30 days prior to enrollment, or prior to receipt of study product, vaccination scab still present; or planned administration within 30 days after enrollment or receipt of study product
* Receipt of any vaccines that are not live attenuated within 14 days prior to enrollment; replication incompetent vaccines such as the Jynneos vaccine for the prevention of monkeypox disease are not considered to be live vaccines
* Receipt of non-HIV experimental vaccine(s) received within the last 1 year. Exceptions may be made by the PSRT for vaccines that have subsequently undergone licensure or Emergency Use Authorization by the FDA or, if outside the United States, by the national regulatory authority or World Health Organization. For volunteers who have received control/placebo in an experimental vaccine trial, the PSRT will determine eligibility on a case-by-case basis
* Initiation of antigen-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval
* Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life greater than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment
* History of serious reaction (eg, hypersensitivity, anaphylaxis) to any related vaccine or component of the study vaccine regimen
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
* Idiopathic urticaria within the past year
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Seizure disorder; febrile seizures as a child or seizures secondary to alcohol withdrawal more than 5 years ago are not exclusionary
* Asplenia or functional asplenia
* Active duty and reserve US military personnel
* Any other chronic or clinically significant condition that in the clinical judgement of the investigator would jeopardize the safety or rights of the study participant, including, but not limited to: clinically significant forms of drug or alcohol abuse, serious psychiatric disorders, persons with any suicide attempt within the past one year (if between 1-2 years, consult PSRT) or cancer that, in the clinical judgment of the site investigator, has a potential for recurrence (excluding basal cell carcinoma)

Asthma is excluded if the participant has ANY of the following:

* Required either oral or parenteral corticosteroids for an exacerbation two or more times within the past year; OR
* Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or co-existing conditions unrelated to asthma); OR
* Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
* Uses medium-to-high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR
* Uses more than one medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than one medication for maintenance therapy daily for greater than two years requires PSRT approval.

  * A participant with a history of an immune-mediated disease, either active or remote. Specific examples are listed in protocol (AESI index). Not exclusionary: 1) remote history of Bell's palsy (>2 years ago) not associated with other neurologic symptoms, 2) mild psoriasis that does not require ongoing systemic treatment
  * Investigator concern for difficulty with venous access based upon clinical history and physical examination. For example, history of IV drug abuse or substantial difficulty with previous blood draws.
  * Presence of implanted electronic medical device (eg, pacemaker, implantable cardioverter defibrillator)
  * Presence of surgical or traumatic metal implant in either upper arm and/or upper torso
  * History of cardiac arrhythmia (eg, supraventricular tachycardia, atrial fibrillation) (Not excluded: sinus arrhythmia)
  * Tattoo overlying the injection sites preventing assessment of reactogenicity in the view of the investigator or skin condition at the injection sites
  * History or presence of keloid scar formation or hypertrophic scar

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - New York Blood Center CRS, New York, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbuilt Vaccine (VV) CRS, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group T1: INO-6160 (2.0 mg) at months 0, 1, 3, 6
- Group T2: INO-6160 (2.0 mg) at months 0, 1, 3, 6 + Trimer-4571 (100 mcg) + 3M-052-AF (5 mcg) + Alum (500 mcg) at months 3, 6
Period: Overall Study
Arm/Group | Group T1 | Group T2
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Reactogenicity symptom | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group T1 | Group T2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 34 [24 to 42] | 30.5 [19 to 45] | 33 [19 to 45]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 | 0 | 0 | 0
  18 - 20 | 0 | 1 | 1
  21 - 30 | 3 | 4 | 7
  31 - 40 | 6 | 4 | 10
  41 - 50 | 1 | 1 | 2
  Above 50 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 7 | 16
  Black or African American | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Multiple Selected | 0 | 3 | 3
  Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Solicited Adverse Events Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured for 14 days after each injection
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Participants
  None | 4 | 0
  Mild | 6 | 7
  Moderate | 0 | 3
  Severe | 0 | 0
  Potentially Life-threatening | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Solicited Adverse Events Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured for 14 days after each injection
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Participants
  Erythema/Redness: None | 4 | 1
  Erythema/Redness: Mild | 4 | 5
  Erythema/Redness: Moderate | 1 | 3
  Erythema/Redness: Severe | 1 | 1
  Erythema/Redness: Potentially Life-threatening | 0 | 0
  Induration/Swelling: None | 8 | 3
  Induration/Swelling: Mild | 1 | 7
  Induration/Swelling: Moderate | 1 | 0
  Induration/Swelling: Severe | 0 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0
  Erythema and/or Induration: None | 4 | 1
  Erythema and/or Induration: Mild | 4 | 5
  Erythema and/or Induration: Moderate | 1 | 3
  Erythema and/or Induration: Severe | 1 | 1
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Solicited Adverse Events Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured for 14 days after each injection
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Participants
  Malaise and/or fatigue: None | 4 | 0
  Malaise and/or fatigue: Mild | 5 | 5
  Malaise and/or fatigue: Moderate | 1 | 4
  Malaise and/or fatigue: Severe | 0 | 1
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0
  Myalgia: None | 8 | 2
  Myalgia: Mild | 1 | 4
  Myalgia: Moderate | 1 | 3
  Myalgia: Severe | 0 | 1
  Myalgia: Potentially Life-threatening | 0 | 0
  Headache: None | 5 | 0
  Headache: Mild | 4 | 6
  Headache: Moderate | 1 | 4
  Headache: Severe | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0
  Nausea: None | 7 | 4
  Nausea: Mild | 3 | 2
  Nausea: Moderate | 0 | 4
  Nausea: Severe | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0
  Chills: None | 9 | 1
  Chills: Mild | 1 | 8
  Chills: Moderate | 0 | 1
  Chills: Severe | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0
  Arthralgia: None | 8 | 5
  Arthralgia: Mild | 1 | 4
  Arthralgia: Moderate | 1 | 1
  Arthralgia: Severe | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0
  Max. Systemic Symptoms: None | 2 | 0
  Max. Systemic Symptoms: Mild | 7 | 1
  Max. Systemic Symptoms: Moderate | 1 | 8
  Max. Systemic Symptoms: Severe | 0 | 1
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0
  Temperature: None | 10 | 6
  Temperature: Mild | 0 | 3
  Temperature: Moderate | 0 | 1
  Temperature: Severe | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0

4. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: The number (percentage) of Participants Reporting Unsolicited Adverse Events (AEs) was summarized by arm
Time Frame: Measured for 30 days after any receipt of study vaccination.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Participants | 6 | 6

5. Primary Outcome: Number of Participants With Early Discontinuation of Vaccinations and Reason for Discontinuation
Description: The number (percentage) of participants with early discontinuation of vaccinations and reason for discontinuation was summarized by arm
Time Frame: Measured through Month 6
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Participants
  Lost to Follow-Up | 1 | 0
  Other | 0 | 1
  Reactogenicity Symptom | 1 | 2
  Did not discontinue SPA | 8 | 7

6. Primary Outcome: Number of Participants With Early Study Termination and Reason for Early Study Termination
Description: The number (percentage) of participants with early study termination and reason for early study termination was summarized by arm
Time Frame: Measured through Month 10
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Participants
  Lost to Follow-Up | 1 | 0
  Reactogenicity Symptom | 0 | 1
  Did not terminate Study | 9 | 9

7. Primary Outcome: Response Rate of Vaccine-matched IgG Binding Antibody (Ab) Responses as Assessed by Multiplex Assay 2 Weeks Following the Fourth Vaccination
Description: The Binding Antibody Multiplex Assay (BAMA) assay was used to evaluate binding antibody responses of each serum specimen against BG505 SOSIP (vaccine trimer immunogen) and Trimer 4571 (vaccine matched immunogen). Positivity criteria include (1) the net Mean Fluorescence Intensity (MFI), or MFI - Blank, values are ≥ antigen-specific cutoff at the 1:50 dilution level for IgG (based on the 95th percentile of the baseline visit serum samples and at least 100 MFI minus Blank), (2) the net MFI values are greater than 3 times the baseline (day 0) net MFI, and (3) the MFI values are greater than 3 times the baseline MFI values. The AB05 antigen was used to assess binding antibody responses to the vaccine-matched trimer INO-6160. The wildtype antigen (BG505 MD39.3) captured both base and non-base specific antibodies, whereas the mutant antigen (BG505 MD39.3-BaseKO), captured only non-base specific antibodies.
Time Frame: Measured at Months 1.5, 3.5, and 6.5
Population: The number of participants with available data after filtering for assay specific quality control criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Participants
  AB05, 1: 50, M1.5 | 1 | 1
  AB05, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  AB05, 1: 50, M3.5 | 5 | 9
  AB05, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  AB05, 1: 50, M6.5 | 5 | 6
  BG505 MD39.3, 1: 50, M1.5 | 7 | 5
  BG505 MD39.3, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  BG505 MD39.3, 1: 50, M3.5 | 8 | 9
  BG505 MD39.3, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  BG505 MD39.3, 1: 50, M6.5 | 8 | 6
  BG505 MD39.3-BaseKO, 1: 50, M1.5 | 1 | 0
  BG505 MD39.3-BaseKO, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  BG505 MD39.3-BaseKO, 1: 50, M3.5 | 4 | 4
  BG505 MD39.3-BaseKO, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  BG505 MD39.3-BaseKO, 1: 50, M6.5 | 4 | 6
  Trimer 4571, 1: 50, M1.5 | 1 | 1
  Trimer 4571, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  Trimer 4571, 1: 50, M3.5 | 4 | 9
  Trimer 4571, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  Trimer 4571, 1: 50, M6.5 | 5 | 6

8. Primary Outcome: Magnitude of Vaccine-matched IgG Binding Antibody (Ab) Responses as Assessed by Multiplex Assay 2 Weeks Following the Third and Fourth Vaccination
Description: The Binding Antibody Multiplex Assay (BAMA) assay was used to evaluate binding antibody responses of each serum specimen against BG505 SOSIP (vaccine trimer immunogen) and Trimer 4571 (vaccine matched immunogen). Epitope specificities are assessed via wildtype-mutant pairs. The AB05 antigen was used to assess binding antibody responses to the vaccine-matched trimer INO-6160. The wildtype antigen (BG505 MD39.3) captured both base and non-base specific antibodies, whereas the mutant antigen (BG505 MD39.3-BaseKO), captured only non-base specific antibodies.
Time Frame: Measured at Months 1.5, 3.5, and 6.5
Population: The number of participants with available data after filtering for assay specific quality control criteria
Measure: Median (Inter-Quartile Range); unit: Net MFI
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Net MFI
  AB05, 1: 50, M1.5 | 72.2 [15.8 to 167.1] | 20.5 [5.4 to 126.4]
  AB05, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  AB05, 1: 50, M3.5 | 484.6 [188.9 to 1241.4] | 3564.5 [1829.2 to 6158.2]
  AB05, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  AB05, 1: 50, M6.5 | 343.9 [196.1 to 1039.7] | 22000 [22000 to 22000]
  BG505 MD39.3, 1: 50, M1.5 | 9633.4 [841.6 to 14037.1] | 2589.8 [433.3 to 12484.8]
  BG505 MD39.3, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  BG505 MD39.3, 1: 50, M3.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000]
  BG505 MD39.3, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  BG505 MD39.3, 1: 50, M6.5 | 22000 [12911.1 to 22000] | 22000 [22000 to 22000]
  BG505 MD39.3-BaseKO, 1: 50, M1.5 | 342.4 [127.3 to 565.6] | 284.5 [122.4 to 699.4]
  BG505 MD39.3-BaseKO, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  BG505 MD39.3-BaseKO, 1: 50, M3.5 | 1266.4 [462.2 to 2177.6] | 1354.5 [501.8 to 3187.5]
  BG505 MD39.3-BaseKO, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  BG505 MD39.3-BaseKO, 1: 50, M6.5 | 1615.9 [655 to 2471.1] | 21943.8 [17194.9 to 22000]
  Trimer 4571, 1: 50, M1.5 | 40.2 [24.6 to 147.6] | 42 [17.6 to 71.8]
  Trimer 4571, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  Trimer 4571, 1: 50, M3.5 | 273.5 [126.8 to 612.2] | 2531.8 [1057.5 to 5427.2]
  Trimer 4571, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  Trimer 4571, 1: 50, M6.5 | 216.8 [77.2 to 605.1] | 22000 [22000 to 22000]

9. Primary Outcome: Response Rate of CD4 + T-cell Responses Measured by Flow Cytometry, to HIV-1-specific Env Peptide Pools, 2 Weeks Following the Third and Fourth Vaccination
Description: Flow cytometry is employed to examine HIV-1-specific CD4+ and CD8+ T-cell responses using a validated Intracellular Cytokine Staining (ICS) assay. To determine positivity, a one-sided Fisher's exact test is applied to a two-by-two contingency table, testing whether the number of cytokine-producing cells for the stimulated data is equal to that for the negative control data.
Time Frame: Measured at Months 3.5 and 6.5
Population: The number of participants with available data after filtering for assay specific quality control criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 8 | 9
Participants
  A-AB05, IFN-g and/or IL-2, M3.5 | 7 | 7
  A-AB05, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  A-AB05, IFN-g and/or IL-2, M6.5 | 8 | 5
  A-AB05, IL-21, M3.5 | 2 | 2
  A-AB05, IL-21, M6.5: number analyzed (Participants) | 8 | 6
  A-AB05, IL-21, M6.5 | 0 | 1
  A-AB05, IL-4 or IL-5 or IL-13 and CD40L, M3.5 | 0 | 0
  A-AB05, IL-4 or IL-5 or IL-13 and CD40L, M6.5: number analyzed (Participants) | 8 | 6
  A-AB05, IL-4 or IL-5 or IL-13 and CD40L, M6.5 | 0 | 0
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M3.5 | 8 | 9
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M6.5 | 8 | 6
  BG505 A-AB05-gp120, IL-21, M3.5 | 2 | 4
  BG505 A-AB05-gp120, IL-21, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp120, IL-21, M6.5 | 0 | 1
  BG505 A-AB05-gp120, IL-4 or IL-5 or IL-13 and CD40L, M3.5 | 0 | 0
  BG505 A-AB05-gp120, IL-4 or IL-5 or IL-13 and CD40L, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp120, IL-4 or IL-5 or IL-13 and CD40L, M6.5 | 0 | 0
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M3.5 | 6 | 9
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M6.5 | 6 | 6
  BG505 A-AB05-gp41, IL-21, M3.5 | 1 | 0
  BG505 A-AB05-gp41, IL-21, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp41, IL-21, M6.5 | 0 | 0
  BG505 A-AB05-gp41, IL-4 or IL-5 or IL-13 and CD40L, M3.5 | 0 | 0
  BG505 A-AB05-gp41, IL-4 or IL-5 or IL-13 and CD40L, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp41, IL-4 or IL-5 or IL-13 and CD40L, M6.5 | 0 | 0
  Total Env, IFN-g and/or IL-2, M3.5 | 8 | 9
  Total Env, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  Total Env, IFN-g and/or IL-2, M6.5 | 8 | 6
  Total Env, IL-21, M3.5 | 2 | 4
  Total Env, IL-21, M6.5: number analyzed (Participants) | 8 | 6
  Total Env, IL-21, M6.5 | 0 | 1
  Total Env, IL-4 or IL-5 or IL-13 and CD40L, M3.5 | 0 | 0
  Total Env, IL-4 or IL-5 or IL-13 and CD40L, M6.5: number analyzed (Participants) | 8 | 6
  Total Env, IL-4 or IL-5 or IL-13 and CD40L, M6.5 | 0 | 0

10. Primary Outcome: Magnitude of CD4 + T-cell Responses Measured by Flow Cytometry, to HIV-1-specific Env Peptide Pools, 2 Weeks Following the Third and Fourth Vaccination
Description: Flow cytometry is employed to examine HIV-1-specific CD4+ and CD8+ T-cell responses using a validated ICS assay
Time Frame: Measured at Months 3.5 and 6.5
Population: The number of participants with available data after filtering for assay specific quality control criteria
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells expressing cytokines
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 8 | 9
% CD4+ T-cells expressing cytokines
  A-AB05, IFN-g and/or IL-2, M3.5 | 0.05 [0.04 to 0.07] | 0.04 [0.02 to 0.08]
  A-AB05, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  A-AB05, IFN-g and/or IL-2, M6.5 | 0.04 [0.04 to 0.06] | 0.06 [0.03 to 0.08]
  A-AB05, IL-21, M3.5 | 0 [0 to 0.02] | 0.01 [0 to 0.01]
  A-AB05, IL-21, M6.5: number analyzed (Participants) | 8 | 6
  A-AB05, IL-21, M6.5 | 0 [0 to 0.01] | 0 [0 to 0.01]
  A-AB05, IL-4 or IL-5 or IL-13 and CD40L, M3.5 | 0 [0 to 0] | 0 [0 to 0]
  A-AB05, IL-4 or IL-5 or IL-13 and CD40L, M6.5: number analyzed (Participants) | 8 | 6
  A-AB05, IL-4 or IL-5 or IL-13 and CD40L, M6.5 | 0 [0 to 0] | 0 [0 to 0]
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M3.5 | 0.14 [0.09 to 0.23] | 0.2 [0.14 to 0.21]
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M6.5 | 0.15 [0.11 to 0.18] | 0.16 [0.15 to 0.17]
  BG505 A-AB05-gp120, IL-21, M3.5 | 0.02 [0.01 to 0.03] | 0.02 [0.02 to 0.03]
  BG505 A-AB05-gp120, IL-21, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp120, IL-21, M6.5 | 0 [0 to 0] | 0.01 [0 to 0.02]
  BG505 A-AB05-gp120, IL-4 or IL-5 or IL-13 and CD40L, M3.5 | 0 [0 to 0] | 0 [0 to 0]
  BG505 A-AB05-gp120, IL-4 or IL-5 or IL-13 and CD40L, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp120, IL-4 or IL-5 or IL-13 and CD40L, M6.5 | 0 [0 to 0] | 0 [0 to 0]
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M3.5 | 0.04 [0.03 to 0.1] | 0.05 [0.04 to 0.07]
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M6.5 | 0.04 [0.03 to 0.05] | 0.05 [0.04 to 0.06]
  BG505 A-AB05-gp41, IL-21, M3.5 | 0.01 [0 to 0.02] | 0.01 [0 to 0.01]
  BG505 A-AB05-gp41, IL-21, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp41, IL-21, M6.5 | 0 [0 to 0] | 0 [0 to 0]
  BG505 A-AB05-gp41, IL-4 or IL-5 or IL-13 and CD40L, M3.5 | 0 [0 to 0] | 0 [0 to 0]
  BG505 A-AB05-gp41, IL-4 or IL-5 or IL-13 and CD40L, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp41, IL-4 or IL-5 or IL-13 and CD40L, M6.5 | 0 [0 to 0] | 0 [0 to 0]
  Total Env, IFN-g and/or IL-2, M3.5 | 0.18 [0.12 to 0.34] | 0.24 [0.18 to 0.32]
  Total Env, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  Total Env, IFN-g and/or IL-2, M6.5 | 0.18 [0.14 to 0.24] | 0.21 [0.21 to 0.22]
  Total Env, IL-21, M3.5 | 0.03 [0.01 to 0.05] | 0.03 [0.02 to 0.03]
  Total Env, IL-21, M6.5: number analyzed (Participants) | 8 | 6
  Total Env, IL-21, M6.5 | 0 [0 to 0] | 0.01 [0 to 0.02]
  Total Env, IL-4 or IL-5 or IL-13 and CD40L, M3.5 | 0 [0 to 0] | 0 [0 to 0]
  Total Env, IL-4 or IL-5 or IL-13 and CD40L, M6.5: number analyzed (Participants) | 8 | 6
  Total Env, IL-4 or IL-5 or IL-13 and CD40L, M6.5 | 0 [0 to 0] | 0 [0 to 0]

11. Primary Outcome: Response Rate of CD8+ T-cell Responses Measured by Flow Cytometry, to HIV-1-specific Env Peptide Pools, 2 Weeks Following the Third and Fourth Vaccination
Description: as for outcome 9
Time Frame: Measured at Months 3.5 and 6.5
Population: The number of participants with available data after filtering for assay specific quality control criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 8 | 9
Participants
  A-AB05, IFN-g and/or IL-2, M3.5 | 1 | 0
  A-AB05, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  A-AB05, IFN-g and/or IL-2, M6.5 | 1 | 0
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M3.5 | 5 | 3
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M6.5 | 5 | 3
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M3.5 | 1 | 0
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M6.5 | 1 | 0
  Total Env, IFN-g and/or IL-2, M3.5 | 6 | 3
  Total Env, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  Total Env, IFN-g and/or IL-2, M6.5 | 6 | 3

12. Primary Outcome: Magnitude of CD8+ T-cell Responses Measured by Flow Cytometry, to HIV-1-specific Env Peptide Pools, 2 Weeks Following the Third and Fourth Vaccination
Description: Flow cytometry is employed to examine HIV-1-specific CD4+ and CD8+ T-cell responses using a validated ICS assay
Time Frame: Measured at Months 3.5 and 6.5
Population: The number of participants with available data after filtering for assay specific quality control criteria
Measure: Median (Inter-Quartile Range); unit: % CD8+ T-cells expressing cytokines
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 8 | 9
% CD8+ T-cells expressing cytokines
  A-AB05, IFN-g and/or IL-2, M3.5 | 0 [0 to 0] | 0 [0 to 0]
  A-AB05, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  A-AB05, IFN-g and/or IL-2, M6.5 | 0 [0 to 0.01] | 0 [0 to 0.01]
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M3.5 | 0.06 [0.01 to 0.15] | 0.02 [0.01 to 0.05]
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp120, IFN-g and/or IL-2, M6.5 | 0.06 [0.02 to 0.19] | 0.06 [0.01 to 0.12]
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M3.5 | 0.01 [0 to 0.01] | 0.01 [0 to 0.02]
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  BG505 A-AB05-gp41, IFN-g and/or IL-2, M6.5 | 0.01 [0 to 0.01] | 0.01 [0 to 0.02]
  Total Env, IFN-g and/or IL-2, M3.5 | 0.11 [0.04 to 0.19] | 0.03 [0.02 to 0.06]
  Total Env, IFN-g and/or IL-2, M6.5: number analyzed (Participants) | 8 | 6
  Total Env, IFN-g and/or IL-2, M6.5 | 0.13 [0.05 to 0.24] | 0.08 [0.02 to 0.14]

13. Secondary Outcome: Neutralizing Ab Magnitude Against Autologous and Tier 1a HIV-1 Isolates as Assessed by TZM-bl Neutralization Assay Following the Third and Fourth Vaccinations
Description: Neutralization assays were used to measure titers in TZM-bl cells against BG505/T332N and MW965.26
Time Frame: Measured at baseline (screening), Month 3.5, and Month 6.5
Population: The number of participants with available data after filtering for assay specific quality control criteria
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Titer
  BG505/T332N, 1: 50, Baseline | 8.2 [5 to 15] | 5 [5 to 10.7]
  BG505/T332N, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  BG505/T332N, 1: 50, M3.5 | 5 [5 to 15.1] | 12.7 [5 to 15.7]
  BG505/T332N, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  BG505/T332N, 1: 50, M6.5 | 5 [5 to 5] | 12.8 [11.2 to 22.1]
  BG505/T332N, 1: 80, Baseline | 5 [5 to 5] | 5 [5 to 5]
  BG505/T332N, 1: 80, M3.5: number analyzed (Participants) | 8 | 9
  BG505/T332N, 1: 80, M3.5 | 5 [5 to 5] | 5 [5 to 5]
  BG505/T332N, 1: 80, M6.5: number analyzed (Participants) | 8 | 6
  BG505/T332N, 1: 80, M6.5 | 5 [5 to 5] | 5 [5 to 5]
  MW965.26, 1: 50, Baseline | 15.9 [13.1 to 19.9] | 16.2 [14.9 to 17.2]
  MW965.26, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  MW965.26, 1: 50, M3.5 | 18.7 [15.6 to 39.3] | 20.1 [16.7 to 34.7]
  MW965.26, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  MW965.26, 1: 50, M6.5 | 23.8 [20.4 to 31.9] | 143.4 [134.7 to 298]
  MW965.26, 1: 80, Baseline | 5 [5 to 5] | 5 [5 to 5]
  MW965.26, 1: 80, M3.5: number analyzed (Participants) | 8 | 9
  MW965.26, 1: 80, M3.5 | 7.8 [5 to 15.7] | 10.9 [5 to 14.2]
  MW965.26, 1: 80, M6.5: number analyzed (Participants) | 8 | 6
  MW965.26, 1: 80, M6.5 | 5 [5 to 10.9] | 47.3 [41.3 to 76.1]
  SVA-MLV, 1: 50, Baseline | 5 [5 to 5] | 5 [5 to 5]
  SVA-MLV, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  SVA-MLV, 1: 50, M3.5 | 5 [5 to 7.8] | 5 [5 to 5]
  SVA-MLV, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  SVA-MLV, 1: 50, M6.5 | 5 [5 to 5] | 5 [5 to 5]
  SVA-MLV, 1: 80, Baseline | 5 [5 to 5] | 5 [5 to 5]
  SVA-MLV, 1: 80, M3.5: number analyzed (Participants) | 8 | 9
  SVA-MLV, 1: 80, M3.5 | 5 [5 to 5] | 5 [5 to 5]
  SVA-MLV, 1: 80, M6.5: number analyzed (Participants) | 8 | 6
  SVA-MLV, 1: 80, M6.5 | 5 [5 to 5] | 5 [5 to 5]

14. Secondary Outcome: Neutralizing Ab Response Rate Against Autologous and Tier 1a HIV-1 Isolates as Assessed by TZM-bl Neutralization Assay Following the Third and Fourth Vaccinations
Description: Neutralization assays were used to measure titers in TZM-bl cells against BG505/T332N and MW965.26. Positivitity call is an unrounded titer >= 10
Time Frame: Measured at baseline (screening), Month 3.5, and Month 6.5
Population: The number of participants with available data after filtering for assay specific quality control criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Participants
  BG505/T332N, 1: 50, Baseline | 5 | 4
  BG505/T332N, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  BG505/T332N, 1: 50, M3.5 | 3 | 5
  BG505/T332N, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  BG505/T332N, 1: 50, M6.5 | 1 | 5
  BG505/T332N, 1: 80, Baseline | 1 | 0
  BG505/T332N, 1: 80, M3.5: number analyzed (Participants) | 8 | 9
  BG505/T332N, 1: 80, M3.5 | 1 | 0
  BG505/T332N, 1: 80, M6.5: number analyzed (Participants) | 8 | 6
  BG505/T332N, 1: 80, M6.5 | 0 | 0
  MW965.26, 1: 50, Baseline | 9 | 10
  MW965.26, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  MW965.26, 1: 50, M3.5 | 8 | 9
  MW965.26, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  MW965.26, 1: 50, M6.5 | 8 | 6
  MW965.26, 1: 80, Baseline | 1 | 0
  MW965.26, 1: 80, M3.5: number analyzed (Participants) | 8 | 9
  MW965.26, 1: 80, M3.5 | 4 | 6
  MW965.26, 1: 80, M6.5: number analyzed (Participants) | 8 | 6
  MW965.26, 1: 80, M6.5 | 3 | 6
  SVA-MLV, 1: 50, Baseline | 2 | 0
  SVA-MLV, 1: 50, M3.5: number analyzed (Participants) | 8 | 9
  SVA-MLV, 1: 50, M3.5 | 2 | 2
  SVA-MLV, 1: 50, M6.5: number analyzed (Participants) | 8 | 6
  SVA-MLV, 1: 50, M6.5 | 1 | 0
  SVA-MLV, 1: 80, Baseline | 1 | 0
  SVA-MLV, 1: 80, M3.5: number analyzed (Participants) | 8 | 9
  SVA-MLV, 1: 80, M3.5 | 0 | 0
  SVA-MLV, 1: 80, M6.5: number analyzed (Participants) | 8 | 6
  SVA-MLV, 1: 80, M6.5 | 0 | 0

15. Secondary Outcome: Differential Binding Response Rates of HIV-1 Specific IgG Binding Ab Responses as Assessed by Multiplex Assay
Description: Epitope specificities are assessed via wildtype-mutant pairs. Serum samples from post-enrollment visits were declared to have positive differential binding responses if they met the following conditions: 1) positive direct binding response, 2) MFI ratio (wild type/mutant type) ≥ 2.5, and wild type at least 250 MFI at selected dilution, 3) net MFI ratio (wild type/mutant type) ≥ 2.5, and wild type at least 250 net MFI at selected dilution. Basespecific binding antibody Area Under the Curve (AUC) values for participants with a positive differential binding response were calculated by subtracting the AUC values of the mutant (BG505-MD39.3 Base-KO untagged) from the AUC values of the wildtype (BG505-MD39.3 untagged)
Time Frame: Measured at Months 1.5, 3.5, and 6.5
Population: The number of participants with available data after filtering for assay specific quality control criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Group T1 | Group T2
Number analyzed (Participants) | 10 | 10
Participants
  BG505_MD39.3_baseKO_1CCv4, 1: 50, M1.5 | 7 | 5
  BG505_MD39.3_baseKO_1CCv4, 1: 250, M3.5: number analyzed (Participants) | 8 | 9
  BG505_MD39.3_baseKO_1CCv4, 1: 250, M3.5 | 8 | 9
  BG505_MD39.3_baseKO_1CCv4, 1: 250, M6.5: number analyzed (Participants) | 8 | 6
  BG505_MD39.3_baseKO_1CCv4, 1: 250, M6.5 | 8 | 4

16. Secondary Outcome: Epitope Specificity of HIV-1 Specific IgG Binding Ab Responses
Description: assessed by multiplex assay
Time Frame: 2 weeks following third vaccination
Reporting Status: Not Posted

17. Secondary Outcome: Response Rate of CD4 +T-cell Responses
Description: measured by flow cytometry, to HIV-1-specific Env peptide pools
Time Frame: 2 weeks following third vaccination
Reporting Status: Not Posted

18. Secondary Outcome: Magnitude of CD4 +T-cell Responses
Description: measured by flow cytometry, to HIV-1-specific Env peptide pools
Time Frame: 2 weeks following third vaccination
Reporting Status: Not Posted

19. Secondary Outcome: Response Rate of CD8+T-cell Responses
Description: measured by flow cytometry, to HIV-1-specific Env peptide pools
Time Frame: 2 weeks following third vaccination
Reporting Status: Not Posted

20. Secondary Outcome: Magnitude of CD8+T-cell Responses
Description: measured by flow cytometry, to HIV-1-specific Env peptide pools
Time Frame: 2 weeks following third vaccination
Reporting Status: Not Posted

21. Secondary Outcome: Magnitude of CD4 +T-cell Responses Measured by Flow Cytometry, to HIV-1-specific Env Peptide Pools
Time Frame: 6 months post last vaccination
Reporting Status: Not Posted

22. Secondary Outcome: Response Rate of CD4 +T-cell Responses Measured by Flow Cytometry, to HIV-1-specific Env Peptide Pools
Time Frame: 6 months post last vaccination
Reporting Status: Not Posted

23. Secondary Outcome: Magnitude of CD8+T-cell Responses Measured by Flow Cytometry, to HIV-1-specific Env Peptide Pools
Time Frame: 6 months post last vaccination
Reporting Status: Not Posted

24. Secondary Outcome: Response Rate of CD8+T-cell Responses Measured by Flow Cytometry, to HIV-1-specific Env Peptide Pools
Time Frame: 6 months post last vaccination
Reporting Status: Not Posted

25. Secondary Outcome: Response Rate of HIV-1 Specific IgG Binding Ab Response
Description: assessed by multiplex assay
Time Frame: 6 months post last vaccination
Reporting Status: Not Posted

26. Secondary Outcome: Magnitude of HIV-1 Specific IgG Binding Ab Response
Description: assessed by multiplex assay
Time Frame: 6 months post last vaccination
Reporting Status: Not Posted

27. Secondary Outcome: Neutralizing Ab Magnitude and Breadth Against Autologous Tier 2 HIV-1 Isolates
Description: assessed by TZM-bl neutralization assay
Time Frame: 6 months post last vaccination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Unsolicited AEs will be collected over a period of 30 days after each vaccination. The Solicited AE assessment were collected through 7 full days after each vaccination.
Arm/Group | Group T1 | Group T2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group T1 (N=10) | Group T2 (N=10)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Solicited) (Gastrointestinal disorders) | 3 (6) | 6 (9)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (Solicited) (General disorders) | 1 (1) | 9 (14)
Fatigue (Solicited) (General disorders) | 6 (12) | 10 (25)
Injection site erythema (Solicited) (General disorders) | 6 (17) | 9 (19)
Injection site pain (Solicited) (General disorders) | 6 (9) | 10 (29)
Injection site swelling (Solicited) (General disorders) | 2 (2) | 7 (9)
Injection site vesicles (General disorders) | 0 (0) | 2 (2)
Anal chlamydia infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Solicited) (Investigations) | 0 (0) | 4 (5)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Solicited) (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (11)
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (17)
Headache (Solicited) (Nervous system disorders) | 5 (8) | 10 (27)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Vulvovaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT05828095/Prot_000.pdf
  • Statistical Analysis Plan: Safety SAP (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT05828095/SAP_001.pdf
  • Statistical Analysis Plan: Immunogenicity SAP (2024-11-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT05828095/SAP_002.pdf